CLINICAL TRIAL: NCT00989560
Title: Post-Operative Crohn's Disease Endoscopic Recurrence "POCER" Study: Endoscopic Guided Therapeutic Intervention & Determination of Cause
Brief Title: Post-operative Crohn's Endoscopic Recurrence Study
Acronym: POCER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Principal Investigator, Michael Kamm, Professorial Fellow, Department of Medicine, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HREC-A 077/09
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active arm (Active Comparator)
  Interventions: Procedure: endoscopy
- Standard care arm (No Intervention)

INTERVENTIONS:
Procedure: endoscopy — patients receive best treatment and care with an additional endoscopy
  Arms: Active arm

SUMMARY:
This randomised, controlled study aims to evaluate the impact of endoscopic assessment, and adjustment of therapy, after surgery in patients with Crohn's disease. The primary endpoint is the severity of endoscopic recurrence. In addition, tissue will be collected for microbiological and immunological analysis.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Crohn's and proven history of disease
* patient undergone surgical resection with creation of a primary anastomosis

Exclusion Criteria:

* endoscopically inaccessible anastomosis by standard colonoscopy
* presence of an end stoma
* pregnancy
* suspected perforation of the gastrointestinal tract
* presence of certain unsuitable comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2009-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Endoscopic recurrence of disease | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Kamm, MBBS MD FRCP FRACP, Principal Investigator — St Vincent's Hospital, Melbourne; University of Melbourne; Peter De Cruz, MBBS, FRACP, Principal Investigator — St Vincent's Hospital, Melbourne; University of Melbourne
Locations (1):
- St Vincent's Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Teh JJ, Berendsen EM, Hoedt EC, Kang S, Zhang J, Zhang F, Liu Q, Hamilton AL, Wilson-O'Brien A, Ching J, Sung JJY, Yu J, Ng SC, Kamm MA, Morrison M. Novel strain-level resolution of Crohn's disease mucosa-associated microbiota via an ex vivo combination of microbe culture and metagenomic sequencing. ISME J. 2021 Nov;15(11):3326-3338. doi: 10.1038/s41396-021-00991-1. Epub 2021 May 25. PMID 34035441
- [Derived] Wright EK, Kamm MA, Dr Cruz P, Hamilton AL, Ritchie KJ, Bell SJ, Brown SJ, Connell WR, Desmond PV, Liew D. Cost-effectiveness of Crohn's disease post-operative care. World J Gastroenterol. 2016 Apr 14;22(14):3860-8. doi: 10.3748/wjg.v22.i14.3860. PMID 27076772
- [Derived] Wright EK, Kamm MA, De Cruz P, Hamilton AL, Ritchie KJ, Krejany EO, Gorelik A, Liew D, Prideaux L, Lawrance IC, Andrews JM, Bampton PA, Sparrow MP, Florin TH, Gibson PR, Debinski H, Gearry RB, Macrae FA, Leong RW, Kronborg I, Radford-Smith G, Selby W, Johnston MJ, Woods R, Elliott PR, Bell SJ, Brown SJ, Connell WR, Desmond PV. Effect of intestinal resection on quality of life in Crohn's disease. J Crohns Colitis. 2015 Jun;9(6):452-62. doi: 10.1093/ecco-jcc/jjv058. Epub 2015 Apr 8. PMID 25855073
- [Derived] Wright EK, Kamm MA, De Cruz P, Hamilton AL, Ritchie KJ, Krejany EO, Leach S, Gorelik A, Liew D, Prideaux L, Lawrance IC, Andrews JM, Bampton PA, Jakobovits SL, Florin TH, Gibson PR, Debinski H, Macrae FA, Samuel D, Kronborg I, Radford-Smith G, Selby W, Johnston MJ, Woods R, Elliott PR, Bell SJ, Brown SJ, Connell WR, Day AS, Desmond PV, Gearry RB. Measurement of fecal calprotectin improves monitoring and detection of recurrence of Crohn's disease after surgery. Gastroenterology. 2015 May;148(5):938-947.e1. doi: 10.1053/j.gastro.2015.01.026. Epub 2015 Jan 22. PMID 25620670
- [Derived] De Cruz P, Kamm MA, Hamilton AL, Ritchie KJ, Krejany EO, Gorelik A, Liew D, Prideaux L, Lawrance IC, Andrews JM, Bampton PA, Gibson PR, Sparrow M, Leong RW, Florin TH, Gearry RB, Radford-Smith G, Macrae FA, Debinski H, Selby W, Kronborg I, Johnston MJ, Woods R, Elliott PR, Bell SJ, Brown SJ, Connell WR, Desmond PV. Crohn's disease management after intestinal resection: a randomised trial. Lancet. 2015 Apr 11;385(9976):1406-17. doi: 10.1016/S0140-6736(14)61908-5. Epub 2014 Dec 24. PMID 25542620